CLINICAL TRIAL: NCT03226067
Title: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Assess the Efficacy & Safety of Oral GKT137831 in Patients With Primary Biliary Cholangitis Receiving Ursodeoxycholic Acid and With Persistently Elevated Alkaline Phosphatase
Brief Title: Study to Assess Safety & Efficacy of GKT137831 in Patients With Primary Biliary Cholangitis Receiving Ursodiol.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSN000300; 2016-004599-23 (EudraCT Number)
Record Dates: First submitted 2017-06-30; First posted 2017-07-21 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-03

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — setanaxib

STUDY DESIGN:
Intervention Model Description: This will be a double-blind, randomized, placebo-controlled, multicenter, parallel group phase 2 trial. A total of 102 subjects will be randomized and allocated to placebo or one of the 2 active treatment arms, according to a 1:1:1 randomization ratio, stratified at study entry by disease severity defined as baseline serum gamma glutamyl transferase (GGT) < 2.5 x ULN or ≥ 2.5 x ULN). Accordingly, approximately 34 subjects will be allocated to each of the 3 treatment arms.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study: the Sponsor, subjects, investigator staff, persons performing the assessments and data reviewers and statisticians will remain blinded to the identity of the study treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GKT137831 400mg twice daily (Experimental): GKT137831 400mg twice daily
  Patients will self-administer 4 capsules in the morning and 4 capsules in the evening.
  Interventions: Drug: GKT137831
- GKT137831 400mg once daily (Experimental): GKT137831 400mg once daily
  Patients will self-administer 4 capsules in the morning and 4 capsules in the evening. The capsules in the evening will be placebos.
  Interventions: Drug: GKT137831; Drug: Placebo oral capsule
- Placebo Arm (Placebo Comparator): Patients will self-administer 4 capsules in the morning and 4 capsules in the evening. All capsules will be placebos.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: GKT137831 — GKT137831 100mg capsules. To be taken as part of two dose arms which are 400mg twice daily or 400mg once daily.
  Other Names: setanaxib
  Arms: GKT137831 400mg once daily; GKT137831 400mg twice daily
Drug: Placebo oral capsule — Matching capsules.
  Other Names: Placebo
  Arms: GKT137831 400mg once daily; Placebo Arm

SUMMARY:
The purpose of this study is to assess the safety and efficacy of GKT13783 in patients with Primary Biliary Cholangitis (PBC) who are taking a stable dose of ursodeoxycholic acid (UDCA) treatment, and have persistently high levels of a liver enzyme called Alkaline Phosphatase (ALP).

DETAILED DESCRIPTION:
Primary biliary cholangitis (PBC) is a disease of the liver. It is caused a sustained attack by the body's immune system on the bile ducts (canals) inside the liver. This continuous assault leads to their gradual destruction and eventual disappearance. This results in obstruction to the flow of bile which gets worse with disease progression. Once the bile duct injury has been established, the disease progresses due to ongoing obstruction of bile flow, inflammation and scarring of the liver tissue(fibrosis). The liver eventually fails.

This research is looking into whether the study drug is better than a dummy drug when given to patients with PBC. This trial will monitor the patients taking part with regular blood tests and ultrasound liver scans before, during, and at the end of the trial. These measures will allow for the ongoing assessment of liver function, and liver stiffness. It is hoped that in patients in whom the study drug is beneficial, the liver function or stiffness may progress at a slower pace, or may even improve during or at the end of the trial. Liver injury, inflammation and fibrosis Participants will be randomly assigned to 1 of 3 treatment groups (active drug once daily, active drug twice daily or placebo). This is a double blinded study so neither the participants nor the staff responsible for their care will know which group they have been assigned to. During the treatment period, participants will take 4 capsules orally at home in the morning and 4 capsules in the evening for 24 weeks.

Participants will be in the trial for 32 weeks in total (about 8 months) and will attend approximately 8 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 80 years, inclusive.
2. Willing and able to give written informed consent and to comply with the requirements of the study.
3. PBC diagnosis as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors:

   * History of elevated ALP levels (> ULN) for at least 6 months
   * Positive anti-mitochondrial antibody (AMA) titer or if AMA negative or in low titer (< 1:80) PBC-specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components [PDC-E2, 2-oxo-glutaric acid dehydrogenase complex])
   * Liver biopsy consistent with PBC (based on historic liver biopsy), including non-suppurative, destructive cholangitis affecting mainly the interlobular and septal bile ducts.
4. Serum ALP ≥ 1.5 x ULN.
5. Serum GGT ≥ 1.5 x ULN.
6. UDCA treatment for at least 6 months and stable dose for at least 3 months prior to Visit 1.
7. Subjects being treated for pruritus with colestyramine must be on a stable dose of colestyramine for at least 8 weeks prior to baseline/Day 1 (Visit 2). Subjects must be willing and able to take colestyramine at least 2 hours before or after study medication.
8. Female subjects of childbearing potential must use a highly effective method of contraception to prevent pregnancy for 4 weeks before randomization and must agree to continue strict contraception for 90 days after last administration of investigational medicinal product (IMP). Male participants with female partners of childbearing potential must be willing to use a condom and require their partner to use an additional form of adequate contraception as approved by the Investigator. This requirement begins at the time of informed consent and ends 90 days after the last administration of IMP. Male study participants must also not donate sperm from baseline until 90 days after the last administration of IMP.

Exclusion Criteria:

1. A positive pregnancy test or breast-feeding for female subjects.
2. Any hepatic decompensation, defined as a past or current history of hepatic encephalopathy, gastrointestinal tract bleeding due to esophageal varices, or ascites.
3. International normalized ratio (INR) > 1.2 unless subject is on anticoagulant therapy.
4. ALT > 3 x ULN.
5. Total bilirubin > 1 x ULN.
6. Planned or current plasmapheresis or other extra-corporeal treatments (e.g., molecular adsorbent recirculation system (MARS)) for treatment-refractory pruritus.
7. History of liver transplantation, current placement on a liver transplant list or current Model for End Stage Liver Disease (MELD) score ≥ 15.
8. Cirrhosis with complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma.
9. Hepatorenal syndrome (type I or II) or Screening serum creatinine > ULN.
10. Competing etiology for liver disease (e.g., hepatitis C, active hepatitis B, non-alcoholic steatohepatitis (NASH), alcoholic liver disease (ALD), autoimmune hepatitis, primary sclerosing cholangitis, Gilbert's Syndrome).
11. Subjects receiving prohibited medications within 3 months of Screening (Visit 1) according to the list (a, b and c) provided in Section 6.6.2.
12. Treatment with any investigational agent within 4 weeks of Visit 1 or 5 half-lives of the investigational medicinal product (whichever is longer).
13. A history of long QT syndrome.
14. Evidence of any of the following cardiac conduction abnormalities during the screening period:

    * A QTc Fredericia interval >450 milliseconds for males and >470 milliseconds for females.
    * A second or third degree atrioventricular block not successfully treated with a pacemaker.
15. History of cancer in the preceding 5 years, except adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, in situ prostate cancer, in situ breast ductal carcinoma, or superficial bladder cancer stage 0).
16. The occurrence of any acute infection requiring systemic antibiotic therapy within the 2 weeks prior the Screening Visit (Visit 1), or human immunodeficiency virus (HIV) infection.
17. A history of bone marrow disorder including aplastic anemia, or marked anemia defined as hemoglobin < 10.0 g/dL (or 6.2 mmol/L).
18. Any condition which, in the opinion of the Investigator, constitutes a risk or contraindication for the participation of the subject in the study, or which could interfere with the study objectives, conduct, or evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Wiesel, MD, Study Director — Calliditas Therapeutics AB
Locations (61):
- United States (21):
  - Mayo Clinic, Phoenix, Arizona
  - University California Davis, Sacramento, California
  - Ventura Clinical Trials, Ventura, California
  - Yale School of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - Jackson Liver and GI Specialist c/o (STAR) LLC, Jackson, Mississippi
  - North Shore University Hospital, Manhasset, New York
  - NYU Hepatology Associates, New York, New York
  - Mount Sinai Health System, New York, New York
  - University of Rochester Medical Centre, Rochester, New York
  - Dayton Gastroenterology Inc., Beavercreek, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - Methodist University Hospital, Memphis, Tennessee
  - St Lukes Episcopal Hospital, Houston, Texas
  - Pinnacle Clinical Research, PLLC, Live Oak, Texas
  - Bon Secours Liver Institute of Hampton Roads, Newport News, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
- Belgium (3):
  - CUB Hôpital Erasme, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (4):
  - University of Calgary Liver Unit, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Centre hospitalier de l'Universite de Montreal (CHUM) Centre de Recherche Service d'Hepatologie, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
- Germany (5):
  - Friedrich-Alexander University Erlangen-Nürnberg, Erlangen, Bavaria
  - Johann Wolfgang Goethe-University, Frankfurt am Main, Hesse
  - Universitatsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mainz, Mainz
- Greece (3):
  - General Hospital of Athens "Hippocratio", Athens
  - Laiko General Hospital, Athens
  - University Hospital of Larissa, Larissa
- Israel (6):
  - Rambam Health Centre, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Centre, Petach-Tiqva
  - Sheba Medical Centre, Ramat Gan
  - Sourasky Tel-Aviv Medical Center, Tel Aviv
- Italy (5):
  - University of Milan-Bicocca, Monza, Lombardy
  - Università Politecnica delle Marche - Facoltà di Medicina e Chirurgia, Ancona
  - Policlinico of Bologna, Bologna
  - San Giovanni Rotondo Hospital (Puglia), Foggia
  - University Hospital Padova, Padua
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Puerta de Hierro-Majadahonda, Madrid
  - University of Alcalá, Madrid
  - Virgen De La Victoria University Hospital, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (9):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Plymouth Hospital NHS Trust, Plymouth, Devon
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, East Yorkshire
  - Gloucestershire Royal Hospital, Gloucester, Gloucestershire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Tayside Medical Science Centre (TASC), Dundee, Tayside
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - King's College Hospital NHS Foundation Trust, London
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Invernizzi P, Carbone M, Jones D, Levy C, Little N, Wiesel P, Nevens F; study investigators. Setanaxib, a first-in-class selective NADPH oxidase 1/4 inhibitor for primary biliary cholangitis: A randomized, placebo-controlled, phase 2 trial. Liver Int. 2023 Jul;43(7):1507-1522. doi: 10.1111/liv.15596. Epub 2023 May 15. PMID 37183520
- [Derived] Jones D, Carbone M, Invernizzi P, Little N, Nevens F, Swain MG, Wiesel P, Levy C. Impact of setanaxib on quality of life outcomes in primary biliary cholangitis in a phase 2 randomized controlled trial. Hepatol Commun. 2023 Feb 20;7(3):e0057. doi: 10.1097/HC9.0000000000000057. eCollection 2023 Mar 1. PMID 36809195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started Sep 2017-Sep 2018
Groups:
- GKT137831 400mg Twice Daily: GKT137831 400mg twice daily
  Patients will self-administer 4 capsules in the morning and 4 capsules in the evening.
  GKT137831: GKT137831 100mg capsules. To be taken as part of two dose arms which are 400mg twice daily or 400mg once daily.
- GKT137831 400mg Once Daily: GKT137831 400mg once daily
  Patients will self-administer 4 capsules in the morning and 4 capsules in the evening. The capsules in the evening will be placebos.
  GKT137831: GKT137831 100mg capsules. To be taken as part of two dose arms which are 400mg twice daily or 400mg once daily.
  Placebo oral capsule: Matching capsules.
Period: Overall Study
Arm/Group | GKT137831 400mg Twice Daily | GKT137831 400mg Once Daily | Placebo Arm
Started | 36 | 38 | 37
Completed | 36 | 38 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GKT137831 400mg Once Daily: Subjects randomized to the 400 mg OD dose arm self-administered IMP twice daily for 24 weeks: 4 active capsules (AM dose) and 4 placebo capsules (PM dose)
- GKT137831 400mg Twice Daily: Subjects randomized to the 400 mg BID dose arm self-administered IMP twice daily for 24 weeks: 4 active capsules (AM dose) and 4 active capsules (PM dose)
- Placebo Arm: Subjects randomized to the placebo arm self-administered placebo twice daily for 24 weeks: 4 placebo capsules (AM dose) and 4 placebo capsules (PM dose)
- Total: Total of all reporting groups
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm | Total
Number analyzed (Participants) | 38 | 36 | 37 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 30 | 91
  >=65 years | 7 | 6 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.1) | 55.6 (9.04) | 56.3 (9.19) | 56.2 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 35 | 99
  Male | 8 | 2 | 2 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 38 | 36 | 36 | 110
  Race: Black | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Greece | 4 | 3 | 3 | 10
  Canada | 3 | 2 | 1 | 6
  Belgium | 5 | 2 | 7 | 14
  United States | 9 | 7 | 11 | 27
  Italy | 5 | 6 | 1 | 12
  United Kingdom | 2 | 8 | 6 | 16
  Israel | 5 | 3 | 5 | 13
  Germany | 2 | 2 | 3 | 7
  Spain | 3 | 3 | 0 | 6
Disease severity level based on baseline serum GGT [Number; unit: participants]
  <2.5 X ULN | 8 | 7 | 10 | 25
  >= 2.5 X ULN | 30 | 29 | 27 | 86

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change in Serum GGT.
Description: Percent change in serum GGT from baseline to Week 24 (serum GGT was measured in U/L)
Time Frame: Baseline to week 24 (visit 7)
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 37 | 30 | 35
percent change | -4.9 (59.58) | -19 (28.89) | -8.4 (21.45)

2. Secondary Outcome: Absolute Change in Serum GGT
Description: Absolute change in serum GGT from baseline to each assessment.
Time Frame: From baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 35 | 37
U/L
  Absolute change W2 | -14.3 (112.66) | -48.5 (61.83) | -11.2 (45.96)
  Absolute change W6 | -22.2 (76.68) | -53.5 (67.57) | -17.9 (59.01)
  Absolute change W12 | -3.9 (115.13) | -50.6 (74.7) | -8.6 (70.11)
  Absolute change W18 | -19.2 (134.32) | -37.9 (93.88) | -4.5 (79.81)
  Absolute change W24 | -17.9 (117.62) | -43.6 (62.22) | -10.7 (78.2)

3. Secondary Outcome: Percent Change in Serum GGT
Description: Percent change in serum GGT from baseline to each assessment (serum GGT was measured in U/L)
Time Frame: From baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 35 | 37
percent change
  Percent change W2 | -7 (25.08) | -17 (17.25) | -6.2 (13.04)
  Percent change W6 | -11.8 (21.59) | -22 (23.4) | -7.5 (16.89)
  Percent change W12 | 1.7 (66.84) | -18.6 (27.44) | -5.5 (19.44)
  Percent change W18 | -4.5 (69.65) | -18.7 (28.55) | -5.2 (22.79)
  Percent change W24 | -4.9 (59.58) | -19 (28.89) | -8.4 (21.45)

4. Secondary Outcome: Percent Change in Serum ALP
Description: Percent change in serum ALP from baseline to each assessment (serum ALP was measured in U/L).
Time Frame: From baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 35 | 37
percent change
  Percent change W2 | -5.5 (10.95) | -13.0 (12.71) | -3.6 (11.51)
  Percent change W6 | -8.6 (13.42) | -16.3 (13.32) | -1.4 (15.19)
  Percent change W12 | -3.9 (22.17) | -14.6 (17.89) | -0.6 (16.41)
  Percent change W18 | -7.8 (21.68) | -15.8 (21.42) | -0.5 (15.66)
  Percent change W24 | -9.7 (21.1) | -12.9 (19.55) | -3.1 (15.99)

5. Secondary Outcome: Absolute Change in Serum ALP
Description: Absolute change in serum ALP from baseline to each assessment.
Time Frame: From baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 35 | 37
U/L
  Absolute change W2 | -19.8 (35.95) | -45.9 (75.75) | -17 (44.4)
  Absolute change W6 | -27.3 (44.13) | -58.6 (63.88) | -14.5 (59.72)
  Absolute change W12 | -15.3 (67.79) | -53 (66.51) | -7.1 (52.75)
  Absolute change W18 | -27.6 (62.54) | -53.2 (80.01) | -6 (50.15)
  Absolute change W24 | -32.5 (65.3) | -45.2 (84.41) | -12.4 (53.48)

6. Secondary Outcome: Absolute Change in Serum Conjugated Bilirubin.
Description: Absolute change in serum conjugated bilirubin from baseline to each assessment.
Time Frame: From baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 32 | 27 | 32
μmol/L
  Absolute change W2 | 0 (1.32) | 0.3 (1.61) | -0.1 (1.4)
  Absolute change W6 | -0.3 (1.14) | 0.5 (2.06) | -0.3 (1.29)
  Absolute change W12 | 0.8 (1.97) | 0.4 (1.28) | -0.1 (1.55)
  Absolue change W18 | 0.5 (2.10) | 0.6 (1.78) | -0.0 (1.91)
  Absolute change W24 | 1.1 (3.44) | 1.1 (1.76) | 0.3 (2.57)

7. Secondary Outcome: Percent Change in Serum Conjugated Bilirubin.
Description: Percent change in serum Conjugated bilirubin, from baseline to each assessment (serum conjugated bilirubin is measured in μmol/L).
Time Frame: From baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 32 | 27 | 32
percent change
  Percent change W2 | 0.9 (16.81) | 5.2 (22.79) | 1.3 (28.11)
  Percent change W6 | -3.4 (18.7) | 6.3 (29.4) | -3.5 (17.99)
  Percent change W12 | 9.4 (27.14) | 4.8 (18.55) | -0.7 (20.81)
  Percent change W18 | 6.0 (28.16) | 8.9 (19.34) | 1.8 (25.98)
  Percent change W24 | 12.7 (36.35) | 16.1 (24.85) | 6.4 (32.90)

8. Secondary Outcome: Absolute Change in Serum Total Bilirubin.
Description: Absolute change in serum total bilirubin, from baseline to each assessment.
Time Frame: from baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 35 | 37
μmol/L
  Absolute change W2 | -0.2 (2.51) | 0.1 (2.76) | -0.4 (3.75)
  Absolute change W6 | -0.5 (2.35) | 0.5 (3.39) | -0.5 (3.29)
  Absolute change W12 | 0.6 (3.35) | 0.1 (2.69) | 0.0 (2.21)
  Absolute change W18 | 0.1 (3.22) | 0.5 (2.82) | -0.1 (3.81)
  Absolute change W24 | 0.5 (3.77) | 1.2 (2.71) | 0.7 (3.23)

9. Secondary Outcome: Percent Change in Serum Total Bilirubin.
Description: Percent change in Serum Total Bilirubin from baseline to each assessment (serum total bilirubin is measured in μmol/L).
Time Frame: from baseline to Weeks 2, 6, 12, 18 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 35 | 37
percent change
  Percent change W2 | -0.6 (23.62) | 5.3 (32.42) | 3.3 (39.98)
  Percent change W6 | -1.6 (21.94) | 8.8 (41.19) | 0.1 (34.6)
  Percent change W12 | 5.7 (32.99) | 7.7 (37.53) | 3.1 (22.39)
  Percent change W18 | 1.7 (28.34) | 9.6 (32.56) | 4.1 (29.5)
  Percent change W24 | 5.4 (29.77) | 14.5 (31.60) | 10.5 (32.27)

10. Secondary Outcome: Absolute Change in Liver Stiffness as Assessed by Transient Elastography (FibroScan® or Similar Technology).
Description: Absolute change in liver stiffness as assessed by transient elastography (FibroScan® or similar technology), from baseline to Week 24, in subjects with values at baseline and Week 24.
Time Frame: From baseline to Week 24, in patients with values at baseline and Week 24.
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 33 | 26 | 32
kPa | -0.5 (5.24) | -0.3 (7.9) | 0.7 (3.63)

11. Secondary Outcome: Percent Change in Liver Stiffness as Assessed by Transient Elastography (FibroScan® or Similar Technology).
Description: Percent change in liver stiffness as assessed by transient elastography (FibroScan® or similar technology), from baseline to Week 24, in subjects with values at baseline and Week 24 (liver stiffness is measured in kPa).
Time Frame: From baseline to Week 24, in patients with values at baseline and Week 24.
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 33 | 26 | 32
percent change | 3.3 (34.95) | 7.9 (43.68) | 10.1 (33.11)

12. Secondary Outcome: Percent Change in Serum Levels of Collagen Fragments Indicative of Collagen Formation and Degradation.
Description: Percent change in serum levels of collagen fragments indicative of collagen formation and degradation, from baseline to Weeks 12 and 24 (serum levels of collagen fragments are measured in ng/mL).
Time Frame: From baseline to Weeks 12 and 24.
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 33 | 34
percent change
  Percent change ProC3 W12 | -2.58 (21.09) | -1.31 (18.23) | 3.64 (27.86)
  Percent change ProC3 W24 | -3.6 (22.54) | 0.69 (18.17) | 3.10 (20.78)
  Percent change ProC5 W12 | 1.17 (20.56) | -6.65 (22.99) | 0.35 (22.52)
  Percent change ProC5 W24 | 2.26 (30.36) | -3.27 (17.73) | -0.51 (37.78)
  Percent change C3M W12 | -0.63 (15.03) | -3.06 (17.73) | 1.31 (20.17)
  Percent change C3M W24 | -0.93 (15.29) | 0.17 (30.10) | -1.06 (23.88)
  Percent change C4M W12 | 1.59 (15.76) | -4.82 (18.97) | 3.19 (20.80)
  Percent change C4M W24 | -4.43 (17.72) | 3.33 (37.63) | 0.73 (21.55)
  Percent change BGM W12 | -0.13 (14.91) | -4.3 (18.81) | -0.12 (23.07)
  Percent change BGM W24 | 1.19 (17.15) | 2.18 (29.14) | 3.77 (25.89)

13. Secondary Outcome: Absolute Change in Liver Stiffness as Assessed by Transient Elastography by Subgroup (FibroScan® or Similar Technology).
Description: Absolute change in liver stiffness by subgroup (>=9.6 kPa) as assessed by transient elastography (FibroScan® or similar technology), from baseline to Week 24, in subjects with values at baseline and Week 24.
Time Frame: From baseline to Week 24, in patients with values at baseline and Week 24.
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 14 | 9 | 16
kPa | -1.9 (7.49) | -2.1 (2.43) | 0.4 (4.65)

14. Secondary Outcome: Percent Change in Liver Stiffness as Assessed by Transient Elastography by Subgroup (FibroScan® or Similar Technology).
Description: Percent change in liver stiffness by subgroup (>=9.6 kPa) as assessed by transient elastography (FibroScan® or similar technology), from baseline to Week 24, in subjects with values at baseline and Week 24 (liver stiffness is measured in kPa).
Time Frame: From baseline to Week 24, in patients with values at baseline and Week 24.
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 14 | 9 | 16
percent change | -5.3 (35.10) | -16.1 (20.71) | 4.2 (30.09)

15. Secondary Outcome: Absolute Change in Pruritis Visual Analogue Scale (VAS) Scores
Description: Absolute Change in Pruritis Visual Analogue Scale (VAS) scores from baseline to weeks 12 and 24- Score from 0 to 10, 0= no itch and 10= severe itch, continuous, day and night intolerable itch.
Time Frame: From baseline to Weeks 12 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 34 | 37
score on a scale
  Absolute change W12 | -0.1 (3.1) | 0.3 (2.33) | 0.5 (1.79)
  Absolute change W24 | -1.0 (2.32) | 0.1 (2.3) | 0.7 (1.83)

16. Secondary Outcome: Percent Change in Pruritis Visual Analogue Scale (VAS) Scores
Description: Percent Change in Pruritis Visual Analogue Scale (VAS) scores from baseline to weeks 12 and 24- Score from 0 to 10, 0= no itch and 10= severe itch, continuous, day and night intolerable itch.
Time Frame: From baseline to Weeks 12 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 34 | 37
percent change
  Percent change W12 | -35.1 (46.13) | -11.7 (73.87) | -8.3 (70.68)
  Percent change W24 | -36.9 (58.6) | -0.3 (92.71) | 27.3 (72.88)

17. Secondary Outcome: Absolute Change in PBC-40 (Primary Biliary Cholongitis) Domain Scores
Description: Absolute Change in PBC-40 Domain scores from baseline to weeks 12 and 24 Symptoms domain: items 1 to 7 of the PBC-40 questionnaire (score from 6 to 35). Itch domain: items 8 to 10 of the PBC-40 questionnaire (score from 0 to 15). Fatigue domain: items 11 to 21 of the PBC-40 questionnaire (score from 11 to 55). Cognitive domain: items 22 to 27 of the PBC-40 questionnaire (score from 6 to 30). Emotional domain: items 28, 30 and 33 of the PBC-40 questionnaire (score from 3 to 15). Social domain: items 29, 31, 32, 34 to 40 of the PBC-40 questionnaire (score from 8 to 50). Higher scores mean worse outcome.
Time Frame: From baseline to Weeks 12 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 34 | 37
score on a scale
  Absolute change Symptoms W12 | -0.4 (3.34) | -0.9 (3.19) | -0.2 (3.52)
  Absolute change Symptoms W24 | 0.1 (3.46) | -1.4 (4.23) | -0.3 (3.10)
  Absolute change Itch W12 | -0.2 (2.61) | 0.6 (2.69) | 0.4 (2.79)
  Absolute change Itch W24 | -0.4 (3.22) | 0.1 (2.83) | 0.1 (2.85)
  Absolute change Fatigue W12 | -1.8 (5.76) | -3.2 (8.25) | 0.6 (4.91)
  Absolute change Fatigue W24 | -0.8 (6.31) | -3.6 (7.32) | 0.6 (5.35)
  Absolute change Cognitive W12 | -0.1 (5.02) | -2.4 (5.68) | 1.0 (4.35)
  Absolute change Cognitive W24 | 0.8 (4.67) | -1.4 (5.34) | 0.3 (3.67)
  Absolute change Emotional W12 | -0.5 (2.09) | -1.8 (3.2) | 0.4 (2.35)
  Absolute change Emotional W24 | -0.3 (2.6) | -2.0 (3.0) | 0.4 (1.78)
  Absolute change Social W12 | 0.6 (4.69) | -2.1 (5.24) | 2.0 (5.43)
  Absolute change Social W24 | 0.8 (5.08) | -2.2 (4.93) | 1.7 (5.01)

18. Secondary Outcome: Percent Change in PBC-40 (Primary Biliary Cholongitis) Domain Scores
Description: Percent Change in PBC-40 Domain scores from baseline to weeks 12 and 24 Symptoms domain: items 1 to 7 of the PBC-40 questionnaire (score from 6 to 35). Itch domain: items 8 to 10 of the PBC-40 questionnaire (score from 0 to 15). Fatigue domain: items 11 to 21 of the PBC-40 questionnaire (score from 11 to 55). Cognitive domain: items 22 to 27 of the PBC-40 questionnaire (score from 6 to 30). Emotional domain: items 28, 30 and 33 of the PBC-40 questionnaire (score from 3 to 15). Social domain: items 29, 31, 32, 34 to 40 of the PBC-40 questionnaire (score from 8 to 50). Higher scores mean worse outcome.
Time Frame: From baseline to Weeks 12 and 24
Population: Number of subjects analyzed in the Intent to Treat population who have evaluable results
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GKT137831 400mg Once Daily | GKT137831 400mg Twice Daily | Placebo Arm
Number analyzed (Participants) | 38 | 34 | 37
percent change
  Percent change Symptoms W12 | -2.8 (24.68) | -2.7 (24.48) | 3.1 (37.21)
  Percent change Symptoms W24 | 1.1 (25.27) | -3.7 (25.19) | 1.1 (35.03)
  Percent change Itch W12 | -5.6 (62.92) | -9.2 (43.43) | -2.5 (48.47)
  Percent change Itch W24 | -11.4 (52.75) | -9.5 (41.83) | -6.8 (40.62)
  Percent change Fatigue W12 | -3.4 (21.11) | -6.8 (26.51) | 3.4 (20.45)
  Percent change Fatigue W24 | 0.3 (24.89) | -9.9 (19.81) | 2.4 (23.07)
  Percent change Cognitive W12 | 6.1 (56.79) | -9.5 (32.14) | 11.7 (51.28)
  Percent change Cognitive W24 | 16.0 (62.27) | -1.9 (40.79) | 5.2 (46.11)
  Percent change Emotional W12 | -1.2 (35.5) | -12.8 (33.88) | 8.7 (45.99)
  Percent change Emotional W24 | 4.9 (54.41) | -16.9 (26.85) | 8.7 (34.49)
  Percent change Social W12 | 4.8 (24.14) | -6.2 (21.65) | 13.9 (40.03)
  Percent change Social W24 | 8.1 (27.94) | -7.7 (18.38) | 9.3 (28.53)

ADVERSE EVENTS:
Time Frame: .Approximately 6-7 months
Description: Adverse events were collected after signing the informed consent form (ICF) and up to completion of the 28-day follow-up period after the last administration of IMP
Arm/Group | GKT137831 400mg Twice Daily | GKT137831 400mg Once Daily | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/38 | 1/37
Other Adverse Events (participants affected / at risk) | 32/36 | 34/38 | 31/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GKT137831 400mg Twice Daily (N=36) | GKT137831 400mg Once Daily (N=38) | Placebo Arm (N=37)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — In the Setanaxib 400 mg BID arm: One (2.8%) subject experienced CTCAE grade 3 multiple fractures, resulting from a road traffic accident.
Urinary Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — One (2.7%) subject in the placebo arm experienced CTCAE grade 1 urinary tract infection. This was considered unrelated to study medication by the investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GKT137831 400mg Twice Daily (N=36) | GKT137831 400mg Once Daily (N=38) | Placebo Arm (N=37)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (3) | 4 (6)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (4) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Gastrooesoghageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (5)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 8 (10) | 8 (11) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Nasopharyngitis (Immune system disorders) | 1 (1) | 3 (3) | 3 (5)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 5 (8) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 5 (8) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3)
Fatigue (General disorders) | 3 (3) | 1 (1) | 8 (8)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 2 (3)
Asthenia (General disorders) | 2 (4) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03226067/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03226067/SAP_003.pdf